CLINICAL TRIAL: NCT00289250
Title: Effect of Antimalarial Treatment on Gametocyte Carriage in Asymptomatic P. Falciparum: A Randomized Controlled Trial
Brief Title: Effect of Antimalarial Treatment on Gametocyte Carriage in Asymptomatic P. Falciparum
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCC867
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2002-12

CONDITIONS: Asymptomatic P.Falciparum Malaria
Keywords: Malaria; Gametocytes; Asymptomatic carriers
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
Drug: Sulfadoxine-pyrimethamine plus artesunate

SUMMARY:
Treatment of uncomplicated P.falciparum malaria with sulfadoxine-pyrimethamine (SP) is followed by a marked increase in the density of gametocytes. To determine whether treatment with SP enhances gametocyte carriage, we randomized asymptomatic carriers of P.falciparum to receive SP alone, SP with a single dose of artesunate, or placebo, and followed them for 56 days to record gametocyte presence and density.

DETAILED DESCRIPTION:
Treatment of P. falciparum malaria with sulfadoxine-pyrimethamine (SP) is followed by a sharp rise in the density of gametocytes. Drug-induced release could enhance transmission of resistant parasites and would argue against the use of SP, especially for intermittent preventive treatment (IPT). We did a randomized trial to determine the effect of treatment with SP on gametocyte carriage. The trial is a three-arm open-label randomized trial. We randomized asymptomatic carriers of P.falciparum to receive antimalarial treatment or placebo, and recorded the prevalence and density of gametocytes over the next 2 months. The trial was conducted during the dry (low malaria transmission) season in four rural villages in The Gambia. Adults and children aged over 6 months who had asexual P.falciparum infection and were confirmed to be free of clinical symptoms of malaria over a 2-day screening period were enrolled and randomized to receive a single dose of SP, or SP plus a single dose of artesunate (SP+AS), or placebo. The primary endpoints were presence of gametocytes 7 and 56 days after treatment, and the duration and density of gametocytaemia over 2 months measured by the area under the curve of gametocyte density against time.

ELIGIBILITY:
Inclusion Criteria:

* P.falciparum parasitaemia above 20/uL
* Resident in one of the four study villages

Exclusion Criteria:

* Fever
* Any other sign of clinical malaria
* Pregnancy
* Weight <5kg
* History of hypersensitivity to any of the study drugs
* Treatment with any of the study drugs in the last 4 weeks

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360
Dates: Start 2001-05; Study Completion 2001-12

PRIMARY OUTCOMES:
Presence of gametocytes 7 days after treatment

SECONDARY OUTCOMES:
Presence of gametocytes 56 days after treatment
Asexual parasitaemia 14 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Pinder, PhD, Study Director — Medical Research Council Unit, The Gambia; Paul J Milligan, PhD, Study Chair — London School of Hygiene and Tropical Medicine; Sam K Dunyo, PhD, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Reseearch Council Laboratories The Gambia, Banjul, The Gambia